CLINICAL TRIAL: NCT07389616
Title: A Clinical Study of Cidabenamine Combined With Azacitidine for Preventing Progression in High-Risk Peripheral T-Cell Lymphoma After Allogeneic Peripheral Blood Hematopoietic Stem Cell Transplantation
Brief Title: A Clinical Trial of Cidabenamine Plus Azacitidine to Prevent Post-Transplant Progression in High-Risk Peripheral T-Cell Lymphoma
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Xianmin Song, MD, Professor, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHSYXY-202503-PTCL
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Peripheral T Cell Lymphoma
Keywords: Peripheral T Cell Lymphoma; Cidabenamine; high-risk; Azacitidine
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cidabenamine combined with Azacitidine (Experimental)
  Interventions: Drug: Cidabenamine, Azacitidine

INTERVENTIONS:
Drug: Cidabenamine, Azacitidine — In the study, Cidabenamine combined with Azacitidine are used as maintenance therapy following allogeneic peripheral blood hematopoietic stem cell transplantation in patients with high-risk peripheral T-cell lymphoma.

SUMMARY:
This study is a single-center, single-arm, prospective, phase II clinical trial designed to evaluate the efficacy and safety of Cidabenamine combined with Azacitidine as maintenance therapy following allogeneic peripheral blood hematopoietic stem cell transplantation in patients with high-risk peripheral T-cell lymphoma.During the screening/baseline period, informed consent will be obtained, and inclusion/exclusion criteria will be verified. The study plans to enroll 40 patients in each group. Enrolled patients will undergo demographic and medical history data collection, along with assessments including vital signs, physical examination, PET-CT, bone marrow aspiration smear, flow cytometry, lymphoid gene rearrangement, and bone marrow pathology.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 70 years, male or female.
2. Diagnosis of peripheral T-cell lymphoma (PTCL) according to the 2022 WHO criteria, including pathological subtypes such as PTCL not otherwise specified (PTCL-NOS), anaplastic large cell lymphoma (ALCL), and angioimmunoblastic T-cell lymphoma (AITL), but excluding hepatosplenic T-cell lymphoma; and meeting at least one of the following high-risk criteria:

   ① Stable Disease (SD) at the time of transplantation;

   ② Relapse after autologous hematopoietic stem cell transplantation (any disease status);

   ③ ≥ Partial Response 1 (PR1).
3. Underwent allogeneic peripheral blood hematopoietic stem cell transplantation for PTCL, with no restriction on donor type.
4. Presence of complete donor chimerism in the bone marrow (T-cell chimerism >95%).
5. ECOG performance status of 0 or 1.
6. Hematological function meeting the following requirements:

   ① Absolute neutrophil count (ANC) ≥ 1.0 × 10⁹/L;

   ② Platelet count (PLT) ≥ 50 × 10⁹/L.
7. Patients must have the ability to understand and be willing to participate in the study and must provide signed informed consent.

Exclusion Criteria:

1. Known hypersensitivity to hypomethylating agents or Cidabenamine.
2. Presence of grade II or higher active acute Graft-versus-Host Disease (GVHD).
3. Presence of moderate or more severe chronic GVHD.
4. Any unstable systemic disease, including but not limited to: unstable angina, cerebrovascular accident or transient ischemic attack (within 3 months prior to screening), myocardial infarction (within 3 months prior to screening), congestive heart failure (New York Heart Association [NYHA] Class ≥ III), status post pacemaker implantation, severe arrhythmia requiring pharmacological treatment, hepatic, renal, or metabolic disease, or pulmonary hypertension.
5. Active, uncontrolled infection, evidenced by any of the following: infection-related hemodynamic instability, worsening or new-onset infectious symptoms/signs, radiologic evidence of a new infectious focus, or persistent fever without localizing symptoms/signs where infection cannot be ruled out.
6. Known HIV infection.
7. Active Hepatitis B (HBV) or active Hepatitis C (HCV) requiring antiviral therapy.
8. History of an autoimmune disease.
9. Pregnant or lactating women.
10. Concurrent participation in another interventional clinical trial and receiving other investigational drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-02-01 (Estimated); Study Completion 2029-08-01 (Estimated)

PRIMARY OUTCOMES:
overall survival (OS) | up to 1 years for the 1y-OS and up to 2 years for the 2y-OS
  The probability of survival at years, measured from the date of transplantation to death from any cause. Patients who are still alive at the time of analysis will be censored on the last follow-up date.

SECONDARY OUTCOMES:
progression-free survival (PFS) | up to 1 years for the 1y-PFS and up to 2 years for the 2y-PFS
  Progression-Free Survival (PFS) is defined as the time from transpalntation until the first occurrence of disease progression or death from any cause, whichever occurs earlier.
non-relapse mortality (NRM) | up to 1 year
  Death occurring after transplantation due to causes other than disease relapse, such as infection, organ toxicity, or transplantation-related complications. Deaths from any cause in the absence of prior relapse are considered events for this endpoint.
cumulative relapse rates (CIR) | up to 1 years for the 1y-CIR and up to 2 years for the 2y-CIR
  The cumulative probability of disease progression (including relapse or progression of the primary disease) within 1 years after transplantation, with non-progression-related death treated as a competing event.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai General hospital,Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No